CLINICAL TRIAL: NCT07184710
Title: Comparative Study Between Methamphetamine Induced Psychosis and Schizophrenia in Sohag Governorate
Brief Title: This Hospital-based Observational Study Employed a Study Will be Conducted in Sohag University Hospital Clinics Aiming to Ensure Cases Presented With Psychosis in Two Phases to Differentiate Into Two Groups a Case of Schizophrenia or a Case of Methamphetamine Induced Psychosis.
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aly Alaa-eldeen Kenawy, M.B.B.Ch_resident in neurology and psychological medicine department_sohag university, Sohag University
Other Study IDs: soh-Med--25-8-3MS
Record Dates: First submitted 2025-09-02; First posted 2025-09-22 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Comparing Clinical Profile and Prognosis of Schizophrenia Versus Methamphetamine Induced Psychosis; SCHIZOPHRENIA; Methamphetamine Induced Psychosis
Keywords: psychosis; schizophrenia; METH; comparative
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months

GROUPS / COHORTS (2):
- schizophrenia
- METH induced psychosis

SUMMARY:
This hospital-based observational study employed prospective follow up study will be conducted in sohag university hospital clinics aiming to ensure cases presented with psychosis in two phases to differentiate into 2 groups (a case of schizophrenia or a case of METH induced psychosis)

Phases-1 includes:

1. Screening and Consent: All consecutive patients meeting initial criteria for psychosis were informed about the study. After explaining the procedures, written informed consent was obtained.
2. Diagnostic Interview: Each participant underwent a SCID-5 interview to confirm DSM-5 diagnoses. The SCID modules relevant to psychotic disorders were used (including the psychotic and substance-use modules). Information from patient self-report and available medical records was incorporated into the diagnostic assessment.
3. Symptom Rating: Following diagnosis, a trained clinician conducted the PANSS interview. This involved structured questions about symptoms over the past week, supplemented by clinical observation. Each PANSS item was scored on a 1-7 scale according to established guidelines. The positive- and negative-symptom subscale scores were recorded for analysis.
4. Clinical Data: A semi-structured form was used to record demographic data, psychiatric history (age at onset, duration of illness), medication history, and details of methamphetamine use (duration, frequency, last use and drug screening). Data were entered into a secure study database.

Phase 2 includes:

Follow up visit after 3 months to obtain :

Positive and Negative Syndrome Scale (PANSS) Drug screening Time of recovery, response to treatment, relapse , job dysfunction duration.

Aim of the study:

The study aims to compare between:

1. Clinical profile-risk factors-of schizophrenia vs methamphetamine induced psychosis in sohag governorate
2. Compare between response to treatment

   * the need of hospitalization and its duration
   * time of recovery
   * job dysfunction duration

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients presenting to the outpatient department with active psychotic symptoms were screened for inclusion. Eligible participants were adults (age ≥18 ≤60) meeting DSM-5 criteria for either methamphetamine-induced psychotic disorder or schizophrenia.

Exclusion Criteria:

* included presence of primary neurological disorders (e.g., epilepsy, dementia), significant medical illness affecting cognition, or inability to participate in interviews.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The sample thus comprised all available patients with methamphetamine-related psychosis or schizophrenia attending the clinic during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-24 (Estimated); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
severity of symptoms of psychosis at time of presentation | from enrollment to 3 Months
  using positive and negative syndrome scale of schizophrenia Positive scale 7 Items, (minimum score = 7, maximum score = 49) includes : Delusions Conceptual disorganization Hallucinations Excitement Grandiosity Suspiciousness/persecution Hostility Negative scale 7 Items, (minimum score = 7, maximum score = 49) includes : Blunted affect Emotional withdrawal Poor rapport Passive/apathetic social withdrawal Difficulty in abstract thinking Lack of spontaneity and flow of conversation Stereotyped thinking General Psychopathology scale 16 Items, (minimum score = 16, maximum score = 112) includes : Somatic concern Anxiety Guilt feelings Tension Mannerisms and posturing Depression Motor retardation Uncooperativeness Unusual thought content Disorientation Poor attention Lack of judgment and insight Disturbance of volition Poor impulse control Preoccupation Active social avoidance PANSS Total score minimum = 30, maximum = 210

SECONDARY OUTCOMES:
improvement after treatment and/or hospitalization | after 3 months of first visit.
  using positive and negative syndrome scale of schizophrenia PANSS Total score minimum = 30, maximum = 210 to compare response to treatment and prognosis of 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Taher abdelrhim Sayed, Prof., Study Chair — faculy of medicine_ sohag university; osama abdelraouf Morad, Ph.D, Study Chair — faculy of medicine_ sohag university; osama eltaher mahmoud, Ph.D, Study Chair — faculy of medicine_ sohag university

IPD SHARING:
Plan to Share IPD: Undecided